CLINICAL TRIAL: NCT02634762
Title: Acute Congestive Heart Failure Urgent Care Evaluation: Prospective Validation of the Emergency Heart Failure Mortality Risk Grade 7-day and 30-day Algorithms in the Emergency Department
Brief Title: Acute Congestive Heart Failure Urgent Care Evaluation
Acronym: ACUTE
Status: Completed | Type: Observational
Sponsor: Institute for Clinical Evaluative Sciences (Other)
Responsible Party: Principal Investigator, Douglas Lee, Senior Scientist, Institute for Clinical Evaluative Sciences
Other Study IDs: 1
Record Dates: First submitted 2015-12-16; First posted 2015-12-18 (Estimated); Last update posted 2018-03-29 (Actual); Status verified 2018-03

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 30 Days
Oversight: Data Monitoring Committee: No

SUMMARY:
This prospective validation study evaluates the ability of a risk algorithm, which can simultaneously predict the risk of death at 7 days and 30 days for patients with acute heart failure presenting to the emergency department. The risk algorithms for prediction of 7-day (Emergency Heart failure Mortality Risk Grade [EHMRG]) and 30-day mortality (EHMRG30-ST) have been previously derived.

ELIGIBILITY:
Inclusion Criteria:

* Patients with acute heart failure diagnosed in the emergency department

Exclusion Criteria:

* Palliative or do-not-resuscitate (DNR) directive
* Dialysis dependent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients presenting to the emergency department diagnosed with heart failure at 8 centers in Ontario, Canada
Sampling Method: Non-Probability Sample
Enrollment: 1983 (Actual)
Dates: Start 2011-01; Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Mortality | 7 days
  Death within 7 days after emergency department presentation for heart failure
Mortality | 30 days
  Death within 30 days after emergency department presentation for heart failure

CONTACTS AND LOCATIONS:
Overall Officials: Douglas Lee, MD, PhD, Principal Investigator — Institute for Clinical Evaluative Sciences
Locations (1):
- University Health Network, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Lee DS, Lee JS, Schull MJ, Borgundvaag B, Edmonds ML, Ivankovic M, McLeod SL, Dreyer JF, Sabbah S, Levy PD, O'Neill T, Chong A, Stukel TA, Austin PC, Tu JV. Prospective Validation of the Emergency Heart Failure Mortality Risk Grade for Acute Heart Failure. Circulation. 2019 Feb 26;139(9):1146-1156. doi: 10.1161/CIRCULATIONAHA.118.035509. PMID 30586748